CLINICAL TRIAL: NCT03002012
Title: Cryptococcal Antigen Screening Plus Sertraline
Acronym: C-ASSERT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: SAEs with n=1 serotonin syndrome, n=2 SAEs after sertraline interruption.
Sponsor: University of Minnesota (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01AI125003 (NIH); U01AI125003 (NIH); 33238 (Other: DAIDS-ES ID)
Record Dates: First submitted 2016-12-14; First posted 2016-12-23 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cryptococcosis; Cryptococcal Infections; AIDS-Related Opportunistic Infections
Keywords: cryptococcal antigen; preemptive treatment; CRAG+; sertraline; fluconazole; randomized clinical trial; HIV
MeSH Terms: conditions — Cryptococcosis; AIDS-Related Opportunistic Infections | interventions — Sertraline; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sertraline (Experimental): Fluconazole Standard of Care + Sertraline
  Interventions: Drug: Sertraline; Drug: Fluconazole
- Control (Placebo Comparator): Fluconazole Standard of Care + Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet; Drug: Fluconazole

INTERVENTIONS:
Drug: Sertraline — sertraline 400mg/day
  Other Names: Zoloft; Lustral; Sertraline hydrochloride
  Arms: Sertraline
Drug: Placebo Oral Tablet — matched placebo tablet
  Other Names: Placebo
  Arms: Control
Drug: Fluconazole — Standard of Care Fluconazole per World Health Organization and Ugandan Guidelines (800mg/day x 2 weeks, 400mg/day x10 weeks, 200mg through 6 months).
  Other Names: Fluconazole 200mg tab

SUMMARY:
Cryptococcal meningitis or "Crypto" is a life threatening fungal infection around the brain that requires hospitalization for treatment for 14 days and then continued therapy. Crypto causes 15-20% of HIV/AIDS-related deaths worldwide. However, this infection can be detected before one develops symptoms and becomes ill. People can be screened for infection by a blood test to detect "cryptococcal antigen," (called CrAg), which is part of the fungus, in blood. The World Health Organization and over 22 countries worldwide recommend CrAg screening of all persons with advanced AIDS entering or re-entering into HIV care.

However, it is not known how best to treat people with cryptococcal antigen in their blood, who don't otherwise yet have symptoms of infection around their brain. If no treatment is given, almost all people will develop infection of the brain and/or die. International guidelines suggest using both HIV medicines and an anti-fungal medicine, called fluconazole, to treat this early infection. However, despite this treatment approximately 1 in 4 people may get sick and/or die.

Researchers have recently discovered another medicine that may work against the Cryptococcus fungus. This medicine is called Sertraline, and it is actually a medicine that has been used for more than 25 years to treat depression (sadness). Sertraline is one of the most commonly used medicines worldwide.

The purpose of this research clinical trial is to determine if standard fluconazole antifungal therapy plus a high dose of Sertraline, will be better than standard fluconazole therapy alone for treating early disseminated cryptococcal infection in persons who are asymptomatic and do not yet have infection of the brain (i.e. meningitis).

This study seeks to test if Sertraline will improve survival through 6-months. Prior studies have shown that >90% of those who survive 6-months will survive >5 years.

DETAILED DESCRIPTION:
This is a double-blind, randomized placebo-controlled clinical trial testing sertraline as an antifungal medicine in combination with fluconazole for treatment of HIV-infected persons with AIDS and asymptomatic cryptococcal antigenemia (CrAg+).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Cryptococcal antigen (CrAg) positive in blood
* Age >=18 years
* Written informed consent
* Women of childbearing potential who are participating in sexual activity that could lead to pregnancy must agree to use one reliable method of contraception while receiving fluconazole >=400mg/day

Exclusion Criteria:

* Prior history of cryptococcal meningitis
* Suspected meningitis or mania
* Suspected/known cirrhosis, jaundice, or alanine aminotransferase (ALT) >5x upper limit of normal
* Receiving an antidepressant medicine
* Receiving antifungal therapy, >1 week
* Pregnant or Breastfeeding
* Contraindication to sertraline or fluconazole
* Current rifampin use or other prohibited medication
* Electrocardiogram corrected QT interval (QTc) >450ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Nalintya, MBChB MPH, Study Director — Infectious Disease Institute; Radha Rajasingham, MD, Study Director — University of Minnesota
Locations (1):
- Infectious Disease Institute, Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
A formal written data sharing plan exists. Protocol and trial documents can be shared. De-identified data can be shared after trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available for at least 5 years
Access Criteria: Upon request to the Principal Investigator

REFERENCES:
- [Result] Boulware DR, Nalintya E, Rajasingham R, Kirumira P, Naluyima R, Turya F, Namanda S, Rutakingirwa MK, Skipper CP, Nikweri Y, Hullsiek KH, Bangdiwala AS, Meya DB. Adjunctive sertraline for asymptomatic cryptococcal antigenemia: A randomized clinical trial. Med Mycol. 2020 Nov 10;58(8):1037-1043. doi: 10.1093/mmy/myaa033. PMID 32415846
- See also: PreventCrypto.org has information and training materials for cryptococcal antigen screening and treatment — http://preventcrypto.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sertraline | Control
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Control | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [26 to 32] | 35 [32 to 38] | 32 [29 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  Uganda | 11 | 11 | 22
On Antiretroviral Therapy (ART) at Radomization [Count of Participants; unit: Participants]
  On ART | 6 | 8 | 14
  Not on ART | 5 | 3 | 8
CD4 Cell Count [Median (Full Range); unit: cells/mm3] | 38 [12 to 86] | 50 [7 to 83] | 42 [7 to 86]

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Meningitis-free Survival
Description: Cryptococcal meningitis free survival with retention-in-care through 6 months
  * Those who die of any cause are failures
  * Those developing symptomatic cryptococcal meningitis are failures
  * Those lost to follow up and unable to be tracked are considered failures
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
Participants | 11 | 9

2. Secondary Outcome: 6-month Survival
Description: Survival through 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
Participants | 11 | 10

3. Secondary Outcome: Cumulative Incidence of Symptomatic Cryptococcal Meningoencephalitis
Description: Cumulative incidence of symptomatic cryptococcal meningoencephalitis through 6 months
Time Frame: 6 months
Measure: Number; unit: meningitis events
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
meningitis events | 0 | 1

4. Secondary Outcome: Number of Clinical Adverse Events (Grade 3-5)
Description: Number of Clinical Adverse Events by Division of AIDS (DAIDS) Scale for Grade 3-5 events through 6 months
Time Frame: 6 months
Measure: Number; unit: number of grade 3-5 adverse events
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
number of grade 3-5 adverse events | 4 | 2

5. Secondary Outcome: Number of Laboratory Grade 3-5 Adverse Events
Description: Number of Laboratory Grade 3-5 Adverse Events through 6 months as per the Division of AIDS (DAIDS) grading scale
Time Frame: 6 months
Measure: Number; unit: number of grade 3-5 adverse events
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
number of grade 3-5 adverse events | 4 | 1

6. Secondary Outcome: All-Cause Premature Study Drug/Placebo Discontinuation
Description: Number of participants whose study drug/placebo use was halted prematurely due to any cause through 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
Participants | 1 | 0

7. Secondary Outcome: Prevalence of Depression by Patient Health Questionnaire (PHQ-9) Over Time
Description: Prevalence of depression by Patient Health Questionnaire (PHQ-9) over 6 months as measured at baseline, 4 weeks, 8 weeks, and 12 weeks. The PHQ-9 is a 9-item instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Items are rated on a scale from 0 (not at all) to 3 (nearly every day). Total score is a sum of 9 item scores (Range 0-27). Greater scores indicate greater depressive symptoms. PHQ-9 scores of: 0-4 Minimal/No depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderate severe depression; 20-27 Severe depression. This endpoint reports the median (interquartile range) of the PHQ-9 scores over time.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
score on a scale
  Week 4 | 5 [2 to 7] | 5 [3 to 7]
  Week 8 | 6 [1 to 9] | 3 [2 to 7]
  Week 12 | 2 [0 to 9] | 2 [0 to 3]

8. Other Pre Specified Outcome: Adherence to Study Drug
Description: Participants' percent adherence to study drug regiment by pharmacy medication counts, representing the percent of the total prescribed medication taken by participants.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: Percent of total prescribed medication t
Arm/Group | Sertraline | Control
Number analyzed (Participants) | 11 | 11
Percent of total prescribed medication t
  Week 2 | 100 [100 to 100] | 100 [96 to 100]
  Week 4 | 100 [94 to 100] | 100 [97 to 100]
  Week 8 | 97 [88 to 100] | 100 [96 to 100]
  Week 12 | 89 [63 to 100] | 100 [100 to 100]

ADVERSE EVENTS:
Time Frame: Through week 24
Arm/Group | Sertraline | Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/11
Serious Adverse Events (participants affected / at risk) | 4/11 | 3/11
Other Adverse Events (participants affected / at risk) | 4/11 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=11) | Control (N=11)
Acute Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mania with Psychotic Disorder (Psychiatric disorders) | 2 (3) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Meningitis (Nervous system disorders) | 0 (0) | 1 (1) — Meningitis complicated by CSF leak
Psychosis with Serotonin Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Death (Infections and infestations) | 0 (0) | 1 (1) — Death due to probable meningitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=11) | Control (N=11)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Leukopenia (Immune system disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Trial was terminated early by the NIAID DSMB for excess harm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03002012/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03002012/SAP_001.pdf